CLINICAL TRIAL: NCT00561574
Title: A Randomized Long-Term Safety Study of Org 50081 in Elderly Outpatients With Chronic Primary Insomnia Examining the Effects of 1.5 mg or 3.0 mg of Org 50081
Brief Title: A Long-Term Safety Study of Org 50081 (Esmirtazapine) in Elderly Outpatients With Chronic Primary Insomnia (176005/P05697/MK-8265-001)
Acronym: Jade
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05697; 176005 (Other: Organon Protocol Number); 2007-003636-35 (EudraCT Number)
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Results first posted 2014-07-07 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Sleep Initiation and Maintenance Disorder; Elderly; Mental Disorder; Dyssomnias; Sleep Disorders; Sleep Disorder, Intrinsic
Keywords: elderly; randomized; double blind
MeSH Terms: conditions — Mental Disorders; Dyssomnias; Sleep Wake Disorders; Sleep Disorders, Intrinsic | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esmirtazapine 1.5 mg (Experimental): Participants receive esmirtazapine 1.5 mg tablets, one tablet administered orally once daily for up to 52 weeks
  Interventions: Drug: Esmirtazapine
- Esmirtazapine 3.0 mg (Experimental): Participants receive esmirtazapine 3.0 mg tablets, one tablet administered orally once daily for up to 52 weeks
  Interventions: Drug: Esmirtazapine

INTERVENTIONS:
Drug: Esmirtazapine — One tablet daily

SUMMARY:
The current study is a 52-week safety study in elderly outpatients with chronic primary insomnia randomized to treatment with 1.5 mg or 3.0 mg of esmirtazapine (Org 50081, SCH 900265, MK-8265) to investigate the safety and tolerability of long-term treatment with esmirtazapine in elderly patients.

DETAILED DESCRIPTION:
Insomnia is a common complaint or disorder throughout the world. About one third of the population in the industrial countries reports difficulty initiating or maintaining sleep, resulting in a non-refreshing or non-restorative sleep. The majority of the insomniacs suffer chronically from their complaints.

The maleic acid salt of Org 4420, code name Org 50081 (esmirtazapine), was selected for development in the treatment of insomnia. The first clinical trial with esmirtazapine was a proof-of-concept trial with a four-way cross-over design. All 3 esmirtazapine dose groups showed a statistically significant positive effect on Total Sleep Time (TST) (objective and subjective) and Wake Time After Sleep Onset (WASO), as compared to placebo.

The current study is a 52-week safety study in elderly outpatients with chronic primary insomnia randomized to treatment with 1.5 mg or 3.0 mg of esmirtazapine to investigate the safety and tolerability of long-term treatment with esmirtazapine in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* are at least 65 years of age at screening;
* sign written informed consent after the scope and nature of the investigation have been explained to them, before screening evaluations;
* are able to speak, read and understand the language of the investigator, study staff (including raters) and the informed consent form, and possess the ability to respond to questions, follow instructions and complete questionnaires;
* have demonstrated capability to independently complete the LogPad questionnaires in the week preceding randomization;
* normal bedtime should be within the 21:00 - 01:00 hour range, with no more variation than 2 hours for 5 nights out of 7;
* have a documented diagnosis of chronic primary insomnia, defined as fulfillment of the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV-TR) criteria for primary insomnia [DSM-IV-TR 307.42]) with a duration of >= 1 month;
* fulfill the following criteria based on medical or sleep history. Each of these criteria should be present for at least 3 nights per week for at least one month;

  * TST <= 6.5 hours
  * WASO >= 60 minutes
  * Sleep Latency (SL) >= 30 minutes

Exclusion Criteria:

* have other sleep disorders (DSM-IV-TR) e.g. rapid eye movement (REM) behavioral disorders, sleep related breathing disorders, periodic leg movement disorder, restless leg syndrome, narcolepsy, circadian sleep wake rhythm disorders, or any parasomnia;
* have any significant medical or DSM-IV-TR psychiatric illness causing the sleep disturbances;
* currently meet diagnostic criteria for DSM-IV-TR depression (Major Depressive Disorder [MDD]) or have been diagnosed and treated for MDD within the last 2 years;
* have signs of dementia or other serious cognitive impairment, defined by a score of less than 26 on the Mini-Mental State Examination (MMSE);
* have a history of bipolar disorder, a history of suicide attempt or a family history of suicide; A family history of suicide is defined as any history of suicide in the first and second degree family (parents, siblings, grandparents, or offspring), or a pattern of completed suicides (more than one) in the third degree family (aunts, uncles, nieces, and nephews);
* are night workers or rotating shift workers;
* are traveling, or have plans to travel, through more than three time zones during the trial, from the screening visit onwards;
* have a significant, unstable medical illness e.g. acute or chronic pain, hepatic, renal, metabolic or cardiac disease;
* have clinically relevant electrocardiogram (ECG) abnormalities at screening, as judged by the investigator;
* have clinically relevant abnormal hematology or biochemistry values at screening, as judged by the investigator;
* have DSM-IV-TR substance abuse or DSM-IV-TR addiction within the last year;
* drink more than 2 alcoholic drinks in a day. One drink is approximately equal to: 12 oz or 360 mL of beer (regular or light), or 4 oz or 120 mL of red or white wine, or 2 oz or 60 mL of desert wine (e.g. port, sherry), or 12 oz or 360 mL of wine cooler (regular or light), or 1 oz or 30 mL or spirits (80 to 100 proof, e.g. whiskey, vodka);
* had serious head injury or stroke within the past year, or a history of (non-febrile) seizures;
* use psychotropic drugs affecting sleep within 2 weeks prior to randomization (fluoxetine: 5 weeks);
* use concomitant medication affecting sleep (see Protocol Section 3.4, Concomitant medication);
* smoke > 15 cigarettes per day and/or can not abstain from smoking during the night;
* drink excessive amounts of caffeinated beverages (more than 500 mg caffeine per day);
* have a positive urine drug screen at screening;
* are routinely sleeping during daytime (napping) for more than 60 minutes per day, 3 times/ week;
* have a body mass index (BMI) >= 36;
* have a known hypersensitivity to mirtazapine or to any of the excipients;
* participated in another clinical trial within the last 30 days prior to screening;
* participated in another clinical trial using esmirtazapine (Org 50081) at any time.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 259 (Actual)
Dates: Start 2008-01-09 (Actual); Primary Completion 2010-02-14 (Actual); Study Completion 2010-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ivgy-May N, Chang Q, Pong A, Winokur A. Esmirtazapine for the treatment of chronic primary insomnia: a randomized long-term safety study in elderly outpatients. J Sleep Med. 2020;17(1):19-30. doi: 10.13078/jsm.190032

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg
Started | 128 | 131
Completed | 80 | 73
Not Completed | 48 | 58
Not completed — Adverse Event | 21 | 24
Not completed — Lack of Efficacy | 11 | 21
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Reason Unrelated to Trial | 6 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Total
Number analyzed (Participants) | 128 | 131 | 259
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.7 (5.2) | 71.1 (5.1) | 70.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 79 | 162
  Male | 45 | 52 | 97

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not related to the study drug.
Time Frame: Up to 53 weeks
Population: The All-Subjects-Treated (AST) population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg
Number analyzed (Participants) | 128 | 131
Participants | 115 | 116

2. Primary Outcome: Number of Participants Who Discontinue Study Drug Due to an AE
Description: as for outcome 1
Time Frame: Up to 52 weeks
Population: The AST population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg
Number analyzed (Participants) | 128 | 131
Participants | 21 | 24

3. Primary Outcome: Change From Baseline in Alertness at Awakening
Description: Alertness at awakening was assessed by participants using a 0-100 mm visual analog scale (VAS) in response to Weekly Sleep Diary question 6 "How did you feel upon awakening over the past 7 days?". Scores could range from 0=Tired to 100=Alert. Baseline was defined as the Day 1 assessment of Days -7 to 1 before any study drug was taken. Change from Baseline was calculated using an observed cases (OC) approach.
Time Frame: Baseline and Week 52
Population: The AST population consisted of all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg
Number analyzed (Participants) | 128 | 131
Score on a Scale
  Baseline (BL) (n=121, 123) | 38.3 (17.2) | 38.3 (18.3)
  Change from BL at Week 52 (n=61, 53) | 25.6 (29.1) | 21.7 (25.1)
Statistical Analysis 1: Comparison: Esmirtazapine 1.5 mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Two-sided significance level of 0.05
Statistical Analysis 2: Comparison: Esmirtazapine 3.0 mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Two-sided significance level of 0.05

4. Primary Outcome: Change From Baseline in Feeling Full of Energy
Description: Feeling full of energy was assessed by participants using a 0-100 mm visual analog scale (VAS) in response to Weekly Sleep Diary question 7 "How full of energy have you felt over the past 7 days?". Scores could range from 0=Terribly tired to 100=Full of energy. Baseline was defined as the Day 1 assessment of Days -7 to 1 before any study drug was taken. Change from Baseline was calculated using an OC approach.
Time Frame: Baseline and Week 52
Population: The AST population consisted of all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg
Number analyzed (Participants) | 128 | 131
Score on a Scale
  BL (n=121, 123) | 42.6 (16.8) | 43.3 (18.2)
  Change from BL at Week 52 (n=61, 53) | 20.1 (29.3) | 20.8 (22.6)
Statistical Analysis 1: Comparison: Esmirtazapine 1.5 mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Two-sided significance level of 0.05
Statistical Analysis 2: Comparison: Esmirtazapine 3.0 mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Two-sided significance level of 0.05

5. Primary Outcome: Change From Baseline in Ability to Work/Function
Description: Ability to work/function was assessed by participants using a 0-100 mm visual analog scale (VAS) in response to Weekly Sleep Diary question 8 "How were you able to work or function over the past 7 days?". Scores could range from 0=Not at all to 100=Very well. Baseline was defined as the Day 1 assessment of Days -7 to 1 before any study drug was taken. Change from Baseline was calculated using an OC approach.
Time Frame: Baseline and Week 52
Population: The AST population consisted of all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg
Number analyzed (Participants) | 128 | 131
Score on a Scale
  BL (n=121, 123) | 46.9 (16.8) | 45.9 (18.7)
  Change from BL at Week 52 (n=61, 53) | 19.7 (27.3) | 21.7 (21.5)
Statistical Analysis 1: Comparison: Esmirtazapine 1.5 mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Two-sided significance level of 0.05
Statistical Analysis 2: Comparison: Esmirtazapine 3.0 mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Two-sided significance level of 0.05

6. Primary Outcome: Change From Baseline in Total Nap Time
Description: Total nap time was assessed by participants in response to Weekly Sleep Diary question 9a "How much time per day did you nap, on average?". Baseline was defined as the Day 1 assessment of Days -7 to 1 before any study drug was taken. Change from Baseline was calculated using an OC approach.
Time Frame: Baseline and Week 52
Population: The AST population consisted of all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg
Number analyzed (Participants) | 128 | 131
Minutes
  BL (n=48, 45) | 23.3 (16.0) | 30.5 (31.6)
  Change from BL at Week 52 (n=18, 14) | 10.7 (65.2) | 2.9 (16.3)
Statistical Analysis 1: Comparison: Esmirtazapine 1.5 mg; Test type: Superiority or Other; p = 0.3129, t-test, 2 sided — Two-sided significance level of 0.05
Statistical Analysis 2: Comparison: Esmirtazapine 3.0 mg; Test type: Superiority or Other; p = 0.3154, t-test, 2 sided — Two-sided significance level of 0.05

7. Secondary Outcome: Change From Baseline in Total Sleep Time (TST)
Description: TST was defined as the time recorded by participants in response to Weekly Sleep Diary question 4 "During the past 7 nights, how much time did you actually spend sleeping, on average?". Baseline was defined as the Day 1 assessment of Days -7 to 1 before any study drug was taken. Change from Baseline was calculated using a last observation carried forward (LOCF) approach.
Time Frame: Baseline and Week 52
Population: The Intent-To-Treat (ITT) population consisted of all participants who received at least one dose of study drug and had at least one postbaseline TST assessment.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg
Number analyzed (Participants) | 128 | 129
Minutes
  BL (n=121,121) | 294.3 (71.0) | 292.3 (67.4)
  Change from BL at Week 52 (n=123,128) | 88.3 (89.5) | 86.3 (96.3)
Statistical Analysis 1: Comparison: Esmirtazapine 1.5 mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Two-sided significance level of 0.05
Statistical Analysis 2: Comparison: Esmirtazapine 3.0 mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Two-sided significance level of 0.05

8. Secondary Outcome: Change From Baseline in Wake Time After Sleep Onset (WASO)
Description: WASO was defined as the time recorded by participants in response to Weekly Sleep Diary question 4 "During the past 7 nights, how much time were you awake, on average, after falling asleep initially?" Baseline was defined as the Day 1 assessment of Days -7 to 1 before any study drug was taken. Change from Baseline was calculated using a LOCF approach.
Time Frame: Baseline and Week 52
Population: The ITT population consisted of all participants who received at least one dose of study drug and had at least one postbaseline WASO assessment.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg
Number analyzed (Participants) | 128 | 129
Minutes
  BL (n=121,121) | 110.2 (88.0) | 102.4 (72.2)
  Change from BL at Week 52 (n=122,128) | -62.7 (81.2) | -47.2 (84.9)
Statistical Analysis 1: Comparison: Esmirtazapine 1.5 mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Two-sided significance level of 0.05
Statistical Analysis 2: Comparison: Esmirtazapine 3.0 mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Two-sided significance level of 0.05

9. Secondary Outcome: Change From Baseline in Sleep Latency (SL)
Description: SL was defined as the time recorded by participants in response to Weekly Sleep Diary question 4 "During the past 7 nights, how long did it take you to fall asleep, on average?" Baseline was defined as the Day 1 assessment of Days -7 to 1 before any study drug was taken. Change from Baseline was calculated using a LOCF approach.
Time Frame: Baseline and Week 52
Population: The ITT population consisted of all participants who received at least one dose of study drug and had at least one postbaseline SL assessment.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg
Number analyzed (Participants) | 128 | 129
Minutes
  BL (n=121,121) | 89.8 (73.6) | 92.5 (79.1)
  Change from BL at Week 52 (n=123,128) | -26.1 (99.2) | -22.2 (101.3)
Statistical Analysis 1: Comparison: Esmirtazapine 1.5 mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Two-sided significance level of 0.05
Statistical Analysis 2: Comparison: Esmirtazapine 3.0 mg; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided — Two-sided significance level of 0.05

10. Secondary Outcome: Change From Baseline in Number of Awakenings (NAW)
Description: NAW was defined as the time recorded by participants in response to Weekly Sleep Diary question 2a "During the past 7 nights, how many times did you wake up, on average?" Baseline was defined as the Day 1 assessment of Days -7 to 1 before any study drug was taken. Change from Baseline was calculated using a LOCF approach.
Time Frame: Baseline and Week 52
Population: The ITT population consisted of all participants who received at least one dose of study drug and had at least one postbaseline NAW assessment.
Measure: Mean (Standard Deviation); unit: Number of Awakenings
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg
Number analyzed (Participants) | 128 | 129
Number of Awakenings
  BL (n=118,114) | 2.5 (1.4) | 2.6 (1.3)
  Change from BL at Week 52 (n=114, 109) | -0.3 (1.3) | -0.4 (1.2)
Statistical Analysis 1: Comparison: Esmirtazapine 1.5 mg; Test type: Superiority or Other; p = 0.0116, t-test, 2 sided — Two-sided significance level of 0.05
Statistical Analysis 2: Comparison: Esmirtazapine 3.0 mg; Test type: Superiority or Other; p = 0.0004, t-test, 2 sided — Two-sided significance level of 0.05

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study drug for serious AEs. Up to 7 days after last dose of study drug for non-serious AEs
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg
Serious Adverse Events (participants affected / at risk) | 9/128 | 6/131
Other Adverse Events (participants affected / at risk) | 83/128 | 102/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine 1.5 mg (N=128) | Esmirtazapine 3.0 mg (N=131)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Narcotic intoxication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine 1.5 mg (N=128) | Esmirtazapine 3.0 mg (N=131)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 9 (9)
Dry mouth (Gastrointestinal disorders) | 10 (13) | 14 (15)
Fatigue (General disorders) | 17 (18) | 15 (18)
Nasopharyngitis (Infections and infestations) | 21 (26) | 17 (21)
Urinary tract infection (Infections and infestations) | 2 (3) | 10 (10)
Weight increased (Investigations) | 11 (13) | 20 (20)
Increased appetite (Metabolism and nutrition disorders) | 5 (7) | 12 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 8 (11)
Dizziness (Nervous system disorders) | 12 (13) | 19 (21)
Headache (Nervous system disorders) | 13 (14) | 12 (13)
Restless legs syndrome (Nervous system disorders) | 3 (3) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 3 (3)
Hypertension (Vascular disorders) | 3 (3) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less